CLINICAL TRIAL: NCT04665037
Title: A Phase 2, Open-Label, Single-Arm, Sequential-Panel Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Posaconazole (POS, MK-5592) Intravenous and Powder for Oral Suspension Formulations in Pediatric Participants From Birth to Less Than 2 Years of Age With Possible, Probable, or Proven Invasive Fungal Infection
Brief Title: Posaconazole (MK-5592) Intravenous and Oral in Children (<2 Years) With Invasive Fungal Infection (MK-5592-127)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5592-127; MK-5592-127 (Other: MSD); PHRR230411-005589 (Registry Identifier: PHRR); 2023-505613-24-00 (Registry Identifier: EU CT); U1111-1292-1190 (Registry Identifier: UTN); 2019-003842-34 (EudraCT Number)
Record Dates: First submitted 2020-12-09; First posted 2020-12-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Invasive Fungal Infection
MeSH Terms: conditions — Invasive Fungal Infections | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Panel A: POS IV (Experimental): Posaconazole 6 mg/kg body weight administered in a single dose by IV infusion on Day 1.
  Interventions: Drug: Posaconazole IV 6 mg/kg
- Panel B: POS IV (Experimental): Posaconazole 6 mg/kg body weight administered twice daily by IV infusion on Day 1, and then once daily from Day 2 to a maximum 84 days.
  Interventions: Drug: Posaconazole IV 6 mg/kg
- Panel B: POS PFS (Experimental): Following a minimum of 7 days IV dosing, participants as clinically able will be transitioned from POS IV to POS PFS nominal 6 mg/kg body weight based on weight bands administered on Day 8, once daily to a maximum 84 days.
  Interventions: Drug: Posaconazole PFS 6 mg/kg

INTERVENTIONS:
Drug: Posaconazole IV 6 mg/kg — POS 6 mg/kg body weight by IV infusion
  Other Names: MK-5592; NOXAFIL®; SCH56592
  Arms: Panel A: POS IV; Panel B: POS IV
Drug: Posaconazole PFS 6 mg/kg — POS nominal 6 mg/kg body weight based on weight bands taken orally
  Other Names: MK-5592; NOXAFIL®; SCH56592
  Arms: Panel B: POS PFS

SUMMARY:
This study aims to estimate the pharmacokinetics (PK) of posaconazole (POS, MK-5592) intravenous (IV) and powder for oral suspension (PFS) formulations in pediatric participants <2 years of age with invasive fungal infection (IFI).

DETAILED DESCRIPTION:
There are 2 panels in this study. In Panel A, POS IV will be evaluated in ≥8 participants. In Panel B, both POS IV and POS PFS will be evaluated in ≥14 participants, including ≥6 who are <3 months of age and ≥5 who transition to the PFS formulation of POS.

ELIGIBILITY:
Inclusion Criteria:

* Panel A: is undergoing treatment for possible, probable, or proven IFI known or suspected to be cause by fungal pathogens against which POS has demonstrated activity (which can include candidiasis)
* Panel B: has an investigator-assessed diagnosis of possible, probable, or proven IFI known or suspected to be cause by fungal pathogens against which POS has demonstrated activity (and cannot include candidiasis)
* Has a central line (eg, central venous catheter, peripherally-inserted central catheter) in place or planned to be in place before beginning IV study intervention.
* Has a body weight of ≥500 g
* The participant (or legally acceptable representative) has provided documented informed consent for the study.

Exclusion Criteria

* Has received POS within 30 days before Day 1
* Has cystic fibrosis, pulmonary sarcoidosis, aspergilloma, or allergic bronchopulmonary aspergillosis
* Has a known hereditary problem of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* Has known or suspected active COVID-19 infection
* Has a known hypersensitivity or other serious adverse reaction to any azole antifungal therapy, or to any other ingredient of the study intervention used
* Has any known history of torsade de pointes, unstable cardiac arrhythmia or proarrhythmic conditions, a history of recent myocardial infarction, congenital or acquired QT interval (QT) prolongation, or cardiomyopathy in the context of cardiac failure within 90 days of first dose of study intervention
* Has received any listed prohibited medications within the specified timeframes before the start of study intervention
* Has a known hereditary problem of galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption (Part B)
* Has suspected/proven invasive candidiasis (Part B)
* Has enrolled previously in the current study and been discontinued
* Has QTc prolongation at screening >500 msec
* Has significant liver dysfunction
* Is hemodynamically unstable, exhibits hemodynamic compromise, or is not expected to survive at least 5 days

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average concentration (Cavg) of single-dose IV POS (Panel A) | Predose, 0.25 and 24 hours post-infusion on Day 1
  The Cavg of IV POS is based on population PK analysis.
Maximum concentration (Cmax) of single-dose IV POS (Panel A) | Predose, 0.25 and 24 hours post-infusion on Day 1
  The Cmax of IV POS is based on population PK analysis.
Time to maximum concentration (Tmax) of single-dose IV POS (Panel A) | Predose, 0.25 and 24 hours post-infusion on Day 1
  The Tmax of IV POS is based on population PK analysis.
Area under the plasma concentration-time curve from dosing to 24 hours postdose (AUC0-24) of single-dose IV POS (Panel A) | Predose, 0.25 and 24 hours post-infusion on Day 1
  The AUC 0-24 of IV POS is based on population PK analysis.
Clearance (CL) of single-dose IV POS (Panel A) | Predose, 0.25 and 24 hours post-infusion on Day 1
  The clearance (CL) of IV POS is based on population PK analysis.
Area under the plasma concentration-time curve from dosing to infinity (AUC0-∞) of single-dose IV POS (Panel A) | Predose, 0.25 and 24 hours post-infusion on Day 1
  The AUC0-∞ of IV POS is based on population PK analysis.
Cavg of multiple-dose IV POS (Panel B) | Predose and 0.25 post-infusion on Day 1; Weeks 1, 2, 4, 6, 9, and 12
  The Cavg of IV POS is based on population PK analysis.
Cmax of multiple-dose IV POS (Panel B) | Predose and 0.25 post-infusion on Day 1; Weeks 1, 2, 4, 6, 9, and 12
  The Cmax of IV POS is based on population PK analysis.
Tmax of multiple-dose IV POS (Panel B) | Predose and 0.25 post-infusion on Day 1; Weeks 1, 2, 4, 6, 9, and 12
  The Tmax of IV POS is based on population PK analysis.
AUC0-24 of multiple-dose IV POS (Panel B) | Predose and 0.25 post-infusion on Day 1; Weeks 1, 2, 4, 6, 9, and 12
  The AUC0-24 of IV POS is based on population PK analysis.
CL of multiple-dose IV POS (Panel B) | Predose and 0.25 post-infusion on Day 1; Weeks 1, 2, 4, 6, 9, and 12
  The CL of IV POS is based on population PK analysis.
Cavg of multiple-dose PFS POS (Panel B) | Predose and 0.25 post-infusion on Day 1; Weeks 1, 2, 4, 6, 9, and 12
  The Cavg of PFS POS is based on population PK analysis.
Cmax of multiple-dose PFS POS (Panel B) | Predose and 0.25 post-infusion on Day 1; Weeks 1, 2, 4, 6, 9, and 12
  The Cmax of PFS POS is based on population PK analysis.
AUC0-24 of multiple-dose PFSPOS (Panel B) | Predose and 0.25 post-infusion on Day 1; Weeks 1, 2, 4, 6, 9, and 12
  The AUC0-24 of PFS POS is based on population PK analysis.

SECONDARY OUTCOMES:
Cavg of IV POS in neonates and infants <2 years of age compared to adults and older pediatric populations (Panel B) | Predose and 0.25 post-infusion on Day 1; Weeks 1, 2, 4, 6, 9, and 12
  The Cavg of IV POS is based on population PK analysis. Comparisons between participants in Panel B will be made to data that was previously collected in older participants.
Percentage of participants with an ≥ 1 adverse event (AE) [Panels A and B] | Up to 98 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants who discontinued study therapy due to an AE (Panels A and B) | Up to 84 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with a drug-related AE (Panels A and B) | Up to 98 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with all-cause mortality (ACM) [Panel B] | Up to 28 days
  The percentage of participants with ACM will be reported.
Percentage of participants with need for systemic antifungal therapy (other than POS) during the study period (Panel B) | Up to 84 days
  Percentage of participants who received additional antifungal therapy in Panel B will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (26):
- United States (5):
  - Rady Children's Hospital-San Diego ( Site 2101), San Diego, California
  - Nicklaus Children's Hospital ( Site 2109), Miami, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago ( Site 2104), Chicago, Illinois
  - Duke University Medical Center ( Site 2106), Durham, North Carolina
  - Driscoll Children's Hospital ( Site 2113), Corpus Christi, Texas
- Belgium (3):
  - UCL Saint Luc ( Site 1050), Brussels, Bruxelles-Capitale, Region de
  - UZ Gent ( Site 1052), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 1051), Leuven, Vlaams-Brabant
- Greece (2):
  - Athens Childrens Hospital Aglaia Kyriakou ( Site 1102), Athens, Attica
  - General Hospital of Thessaloniki "Ippokrateio" ( Site 1100), Thessaloniki
- Israel (4):
  - Rambam Medical Center ( Site 1402), Haifa
  - Hadassah Ein Karem Hebrew University Medical Center ( Site 1401), Jerusalem
  - Sheba Medical Center ( Site 1404), Ramat Gan
  - Sourasky Medical Center ( Site 1403), Tel Aviv
- Mexico (3):
  - Instituto Nacional de Pediatria-Unidad de Apoyo a la Investigación Clínica ( Site 2200), Mexico City, Mexico City
  - Hospital Infantil de Mexico Federico Gomez-Infectious Diseases ( Site 2202), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Infectologia ( Site 2203), Monterrey, Nuevo León
- Instituto Nacional de Enfermedades Neoplasicas ( Site 1601), Lima, Peru
- Poland (2):
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckieg-Klinika Transplantacji Szpiku, Onkolog ( Site 1708), Wroclaw, Lower Silesian Voivodeship
  - Wojewodzki Specjalistyczny Szpital Dzieciecy ( Site 1705), Olsztyn, Warmian-Masurian Voivodeship
- Russia (3):
  - Mechnikov State Medical University ( Site 1803), Saint Petersburg, Sankt-Peterburg
  - Pavlov State Medical University ( Site 1801), Saint Petersburg, Sankt-Peterburg
  - Regional Children Clinical Hospital 1 ( Site 1802), Yekaterinburg, Sverdlovsk Oblast
- Seoul National University Hospital-Pediatrics ( Site 2600), Seoul, South Korea
- Ukraine (2):
  - Ivano-Frankivsk Regional Pediatric Clinical Hospital ( Site 1911), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - NATIONAL CHILDREN'S SPECIALIZED HOSPITAL "OKHMATDYT" OF THE -Intensive Care Unit ( Site 1912), Kiev, Kyiv Oblast

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26165&tenant=MT_MSD_9011